CLINICAL TRIAL: NCT03169465
Title: Open Versus Endoscopic Surgical Management Of Posterior Calcaneal (HAGLUND) Deformity. A Pilot Non Randomized Trial
Brief Title: Open Versus Endoscopic Surgical Management Of Posterior Calcaneal Deformity.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, MAHassan, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCD
Record Dates: First submitted 2017-05-25; First posted 2017-05-30 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Bone Diseases
MeSH Terms: conditions — Bone Diseases | interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- open group (Experimental): patients with posterior calcaneal deformity
  Interventions: Procedure: open approach
- endoscopic group (Active Comparator): patients with posterior calcaneal deformity
  Interventions: Procedure: endoscopic approach

INTERVENTIONS:
Procedure: open approach — open excision of the bursa and deformity then debridement of Achilles tendon
  Arms: open group
Procedure: endoscopic approach — excision of the bursa and deformity then debridement of Achilles tendon through endoscopy
  Arms: endoscopic group

SUMMARY:
Patients with posterior calcaneal deformity may presented by many clinical data associated with retrocalcaneal bursitis which occurs due to the deformity this clinical complaining include pain and swelling in the back of the heel.

Many treatment choices available of this deformity with low level of response to conservative treatment which includes medical treatment , physiotherapy and corticosteroids injection. surgical treatment in cases of HAGLUND deformity is the treatment of choice including either endoscopic or open surgical approach for this deformity .

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic patients.
* Continued refractory pain despite use of extensive conservative management.

Exclusion Criteria:

* Asymptomatic patients
* Patients which are unfit for surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2018-05 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
the mean difference in pain scores postoperative | 3 months
  visual analog scale

IPD SHARING:
Plan to Share IPD: No